CLINICAL TRIAL: NCT05064670
Title: EX-MED Cancer Sweden: A Randomised Controlled Trial of Distance-based Exercise for People Treated for Cancer
Brief Title: Exercise as Medicine for People With Cancer Sweden
Acronym: EX-MED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Cancer Society (Other); SATS (Unknown)
Responsible Party: Principal Investigator, Yvonne Wengstrom, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2019-04151
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer; Breast Cancer; Colorectal Cancer
Keywords: Exercise; Cancer; Fitness; Distance-based; Home-based
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The intervention group will, in addition to routine clinical care according to (inter-) national guidelines, receive an exercise program of resistance and aerobic exercise delivered live online by an upskilled exercise professional in group exercise classes twice weekly for 3 months
  Interventions: Behavioral: Exercise
- Control (No Intervention): The control group will receive routine clinical care according to (inter-) national guidelines

INTERVENTIONS:
Behavioral: Exercise — A twice weekly, 3-month supervised exercise program of whole body resistance training using body weight and a resistance band, and moderate to high intensity aerobic activities, consisting of a consecutive series of timed exercises performed one after the other (14-18 on the Borg scale). Classes are conducted live in groups through Microsoft Teams. Participants will not receive any contact or exercise support in the 3-month follow-up period following the initial 3-month intervention
  Arms: Exercise

SUMMARY:
Regular exercise has been shown to have beneficial health effects in cancer survivors, including improving quality of life and other important health outcomes. However, providing people with cancer with easily accessible, high-quality exercise support and programs is a challenge. Therefore, there is a need to develop easily accessible exercise programs that draw upon the current evidence. Supervised, distance-based exercise programs have the benefit of reaching out to many people while providing the support of an exercise professional.

The aim of the EX-MED Cancer Sweden trial is to examine the effectiveness of a supervised, distance-based exercise program, in people previously treated for breast, prostate, or colorectal cancer, on health-related quality of life (HRQoL), as well as other physiological and patient-reported health outcomes. Participants will be randomized to a 3-month supervised, distance-based exercise program or to a usual care control group.

Testing timepoints are baseline, 3 months (end of intervention) and 6 months (3 month followup). At these timepoints, patients will be asked to fill in online questionaires, and and undergo physical tests. A selection of the particpants and personal trainers involved in the intervention will also be invited to participate in focus group discussion or interviews about the experiences of being involved in the EX-MED Cancer Sweden program.

DETAILED DESCRIPTION:
The primary aim of the study is to examine the effectiveness of EX-MED Cancer Sweden on health-related quality of life in people diagnosed with breast, prostate, and colorectal cancer.

The secondary aims are to examine the effect of the program on other important endpoints such as physical activity level, physical function, muscle strength, exercise capacity, symptoms, and body composition (lean and fat mass).

To determine the sustainability of the effects of the supervised program, the study includes a 3-month follow-up time point (6 months post-baseline)

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* males or females
* people diagnosed with any type of stage I-IIIa breast, prostate or colorectal cancer who have undergone and completed curative treatment (note: participants are eligible if they are currently receiving/scheduled to receive anti-hormonal therapy) at the Karolinska Comprehensive Cancer Centre, Sweden

Exclusion Criteria:

* currently receiving or scheduled to receive cancer treatment (except anti-hormonal therapy)
* any medical conditions that may prevent safe participation in the testing or exercise demands of the study
* performing regular exercise throughout the last month defined as undertaking at least 150 mins moderate intensity aerobic exercise and two or more structured resistance exercise sessions per week
* unable to read and speak Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Baseline, 3 months
  Assessed by the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) (global quality of life summary scale). Patients responds to questions about their quality of life on a scale of 1- (not at all) to 4 (alot).
Health-related quality of life | 3 months
  Assessed by the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) (global quality of life summary scale). Patients responds to questions about their quality of life on a scale of 1- (not at all) to 4 (alot).

SECONDARY OUTCOMES:
Cancer related fatigue | Baseline
  Assessed by the Piper Fatigue scale (PFS) (total cancer related fatigue scale). Participants respond to questions about their fatigue on a scale of 1 (being positive)-10 (being bad/negative)
Cancer related fatigue | 3 months
  Assessed by the Piper Fatigue scale (PFS) (total cancer related fatigue scale). Participants respond to questions about their fatigue on a scale of 1 (being positive)-10 (being bad/negative)
Cancer related fatigue | 6 months
  Assessed by the Piper Fatigue scale (PFS) (total cancer related fatigue scale). Participants respond to questions about their fatigue on a scale of 1 (being positive)-10 (being bad/negative)
Symptoms and symptom burden (total symptoms scale) | Baseline
  Assessed by the memorial symptom assessment scale (MSAS) (total symptoms scale). Patients respond to how often the have had the symptoms (1-almost never- 4 almost always), how severe the symptoms have been (1- light - 4- very severe) and how distressing the symptoms were to them (0- not at all- to 4 very)
Symptoms and symptom burden (total symptoms scale) | 3 months
  Assessed by the memorial symptom assessment scale (MSAS) (total symptoms scale). Patients respond to how often the have had the symptoms (1-almost never- 4 almost always), how severe the symptoms have been (1- light - 4- very severe) and how distressing the symptoms were to them (0- not at all- to 4 very)
Symptoms and symptom burden (total symptoms scale) | 6 months
  Assessed by the memorial symptom assessment scale (MSAS) (total symptoms scale). Patients respond to how often the have had the symptoms (1-almost never- 4 almost always), how severe the symptoms have been (1- light - 4- very severe) and how distressing the symptoms were to them (0- not at all- to 4 very)
Cardiorespiratory fitness | Baseline
  Estimated/predicted maximal oxygen uptake, VO2max assessed by the Ekblom-Bak submaximal cycle test
Cardiorespiratory fitness | 3 months
  Estimated/predicted maximal oxygen uptake, VO2max assessed by the Ekblom-Bak submaximal cycle test
Cardiorespiratory fitness | 6 months
  Estimated/predicted maximal oxygen uptake, VO2max assessed by the Ekblom-Bak submaximal cycle test
Physical function of the lower body | Baseline
  Assessed by the 5 sit to stand test (seconds)
Physical function of the lower body | 3 months
  Assessed by the 5 sit to stand test (seconds)
Physical function of the lower body | 6 months
  Assessed by the 5 sit to stand test (seconds)
Upper body muscle strength | Baseline
  Assessed by a hypothetical 12-RM chest press test
Upper body muscle strength | 3 months
  Assessed by a hypothetical 12-RM chest press test
Upper body muscle strength | 6 months
  Assessed by a hypothetical 12-RM chest press test
Lower body muscle strength | Baseline
  Assessed by a hypothetical 12-RM leg press test
Lower body muscle strength | 3 months
  Assessed by a hypothetical 12-RM leg press test
Lower body muscle strength | 6 months
  Assessed by a hypothetical 12-RM leg press test
Whole body muscle mass | Baseline
  Assessed by bio impendence device (InBody770) (kg)
Whole body muscle mass | 3 months
  Assessed by bio impendence device (InBody770) (kg)
Whole body fat mass | 6 months
  Assessed by bio impendence device (InBody770) (kg)
Whole body fat percentage | Baseline
  Assessed by bio impendence device (InBody770) (%)
Whole body fat percentage | 3 months
  Assessed by bio impendence device (InBody770) (%)
Whole body fat percentage | 6 months
  Assessed by bio impendence device (InBody770) (%)
Self reported physical activity | Baseline
  Assessed by the Godin Leisure time physical activity questionnaire (mins). Patients detail how many minutes per week they have performed vigorous, moderate and low intensity physical activity
Self reported physical activity | 3 months
  Assessed by the Godin Leisure time physical activity questionnaire (mins). Patients detail how many minutes per week they have performed vigorous, moderate and low intensity physical activity
Self reported physical activity | 6 months
  Assessed by the Godin Leisure time physical activity questionnaire (mins). Patients detail how many minutes per week they have performed vigorous, moderate and low intensity physical activity
Self efficacy of exercise | Baseline
  Assessed by the Self-Efficacy of Exercise (SEE) questionnaire (total score). Patients respond to questions ranging from 0 (not at all sure) to 10 (completely sure)
Self efficacy of exercise | 3 months
  Assessed by the Self-Efficacy of Exercise (SEE) questionnaire (total score). Patients respond to questions ranging from 0 (not at all sure) to 10 (completely sure)
Self efficacy of exercise | 6 months
  Assessed by the Self-Efficacy of Exercise (SEE) questionnaire (total score). Patients respond to questions ranging from 0 (not at all sure) to 10 (completely sure)
Quality adjusted life years | Baseline
  Assessed by the EQ-5D-5L questionnaire . Patients rate their health from 0 (worst health you can imagine)-100 (best health you can imagine)
Quality adjusted life years | 3 months
  Assessed by the EQ-5D-5L questionnaire . Patients rate their health from 0 (worst health you can imagine)-100 (best health you can imagine)
Quality adjusted life years | 6 months
  Assessed by the EQ-5D-5L questionnaire . Patients rate their health from 0 (worst health you can imagine)-100 (best health you can imagine)
Health-related quality of life | 6 months
  Assessed by the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) (global quality of life summary scale). Patients responds to questions about their quality of life on a scale of 1- (not at all) to 4 (alot).

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Wengström, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institute/ Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be stored via the Swedish National Data Service (SND) and provided a Digital Object Identifier (DOI).SND is a trusted digital repository, certified against CoreTrustSeal. Through their system DORIS, an examination of the metadata quality carried out by the KI Data Access Unit will be conducted of the data. When the data description is complete, it is published in the SND research data catalog.
Supporting Information: Analytic Code
Time Frame: The data will become available within 5 years of study completion and will be available for visibility and accessibility for 10 years.
Access Criteria: Researchers will have to apply through SND using DORIS to access the data. Once approved, the data is released.

REFERENCES:
- [Derived] Kotte M, Bolam KA, Altena R, Cormie P, Wengstrom Y, Mijwel S. Effects of live-remote exercise on quality of life and other health-related outcomes in cancer survivors: a randomised controlled trial. J Cancer Surviv. 2025 Jun 5. doi: 10.1007/s11764-025-01845-x. Online ahead of print. PMID 40467967
- [Derived] Kotte M, Bolam KA, Mijwel S, Altena R, Cormie P, Wengstrom Y. Distance-based delivery of exercise for people treated for breast, prostate or colorectal cancer: a study protocol for a randomised controlled trial of EX-MED Cancer Sweden. Trials. 2023 Feb 17;24(1):116. doi: 10.1186/s13063-023-07152-z. PMID 36800978